CLINICAL TRIAL: NCT07151482
Title: Impact of Oral Supplementation With Bioactive Collagen Peptides and Other Functional Ingredients on Quality of Life, Related to Vaginal Atrophy and Urinary Incontinence Inwomen With Genitourinary Syndrome of Menopause (GSM)
Brief Title: Impact of Oral Supplementation With Bioactive Collagen Peptides and Other Functional Ingredients
Acronym: Maicol
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7441
Record Dates: First submitted 2025-07-02; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Genitourinary Syndrome of Menopause

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Collagendep — The purpose of this study is to evaluate the improvement of quality of life, vulvovaginal atrophy (VVA) and of initial Urinary Incontinence (UI) in menopausal women with GSM symptoms following oral administration of a food supplement treatment containing 2.5 g of BCP® and other functional ingredients taken once daily over a period of 16 weeks.
  Other Names: QOL questionnaires

SUMMARY:
Genitourinary Syndrome of Menopause (GSM), characterized by vaginal dryness, pain, urinary incontinence, and other symptoms, can be mitigated through both hormonal and non-hormonal treatments. Collagen peptides have shown promising results in improving skin, cartilage, and exhibiting antioxidative activities in studies. This study evaluates changes of quality of life and sexual function, related to vulvovaginal atrophy (VVA) and initial urinary incontinence (UI) in women with GSM symptoms, with the intake of a daily oral food supplement containing 2.5 g of Bioactive Collagen Peptides (BCP®) and other functional ingredients over a 16-week period . This can represent a new therapeutic option for these patients, particularly when hormonal therapy is not an option.

DETAILED DESCRIPTION:
Genitourinary Syndrome of Menopause (GSM) includes a variety of symptoms related to the decline of circulating ovarian hormones. The syndrome is characterized by complaints of vaginal dryness, dyspareunia, pain, urinary incontinence, and recurrent urinary tract infections.

Collagen hydrolysate (CH) has been used in pharmaceuticals and food supplements for improving skin and cartilage tissues. It is absorbed in the digestive tract, appears in the human blood partly in a small peptide form. Based on in vitro studies, collagen peptides (CPs) have shown to exert potent antioxidative activities in different oxidative systems.

The purpose of this study is to evaluate the improvement of quality of life, vulvovaginal atrophy (VVA) and of initial Urinary Incontinence (UI) in menopausal women with GSM symptoms following oral administration of a food supplement treatment containing 2.5 g of BCP® and other functional ingredients taken once daily over a period of 16 weeks. The improvement of systemic health state and satisfaction with this supplement will be evaluated using both subjective and objective measures.

The aim is also to identify significant improvement in quality of sexual function and health of genitourinary system.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal women (at least 12 months since last menstrual period or bilateral oophorectomy)
* Patients with Genitourinary Syndrome and the presence of vulvovaginal atrophy/vestibular trophism alteration (defined as Vaginal Health Index - VHI - less than 15; and Vestibular Trophic Health Score - VeTH - more than 5) and/or initial urinary incontinence based on patient history (stress incontinence , urge incontinence, nicturia reported by patients,) positive IU tests (Stamey score 1: loss of urine with sudden increase in abdominal pressure such as from coughing, sneezing, or laughing) and on a standardized stress test provocation [(cough test supine and in a standing position with a full bladder (300 ml)] in healthy post-menopausal women and/or positive OABSS score for overactive bladder.
* Patients willing to provide Informed consent to participate in the study.
* Women aged between 45 and 65 years.

Exclusion Criteria:

* Renal insufficiency or sever nephropathy.
* In case of known hypersensitivity to one or more of the components contained in the food supplement.
* Active or recent (30 days) genitourinary tract infection.
* Abnormal uterine bleeding.
* Use of lubricants or any other local or systemic preparations, within the 30 days prior to the study.
* Genital prolapse (grade II - III according to the Pelvic Organ Prolapse-Quantification, POP-Q, system classification).
* Serious or chronic condition that could interfere with study compliance.
* Treatment with hormones or other medicines to relieve menopausal symptoms within the 3 months prior the study.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Menopausal women (at least 12 months since last menstrual period or bilateral oophorectomy). Patients with Genitourinary Syndrome in particular suffering of vaginal dryness and/or urinary incontinence.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Quality of life in patient with GSM | 24 weeks
  Evaluate the improvement of quality of life in relation to genitourinary symptoms, to evaluate acceptability and satisfaction with the use of collagen oral supplement in the treatment of Genitourinary Syndrome of Menopause (GSM).
  Quality of life will be evaluate through: QUOL questionnaire SF-12 (during visit T0 and T3). It's a 12-item questionnaire used to assess generic health outcomes from the patient's perspective like: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health.
Sexual function in patient with GSM | 24 weeks
  Evaluate the improvement of sexual function in relation to genitourinary symptoms, to evaluate acceptability and satisfaction with the use of collagen oral supplement in the treatment of Genitourinary Syndrome of Menopause (GSM) with:
  - Female Sexual Function Index (FSFI - short form). FSFI has 19-item and includes: desire (2 items), arousal (4 items), lubrication (4 items), orgasm (3 items), satisfaction (3 items), and pain (3 items). The score scale range is from 0 (worse) to 30 (better score)

SECONDARY OUTCOMES:
Evaluation of vaginal symptoms (included in genitourinary symptoms) | 24 weeks
  Evaluation of genitourinary symptoms (which include both vaginal symptoms and urinary incontinence symptoms).
  vaginal symptoms will be performed using the following tool:
  - Visual Analog Scale (VAS) for the severity of atrophy symptoms (pain, dryness, irritation and leucorrhea), score 0 (better) - 10 (worse).
Evaluation of urinary symptoms (included in genitourinary symptoms) | 24 weeks
  Evaluation of genitourinary symptoms (which include both vaginal symptoms and urinary incontinence symptoms).
  urinary symptoms will be performed using the following tool:
  - International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) where maximum score of 21 represents permanent incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Villa, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS